CLINICAL TRIAL: NCT06267131
Title: Transcutaneous Pulse Oximetry Brain Monitoring Study (US): T-POT Study
Brief Title: Transcutaneous Pulse Oximetry Brain Monitoring Study (US)
Acronym: T-POT US
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cyban Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 22-1286
Record Dates: First submitted 2023-11-08; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Acute Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Single center prospective observational cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled patients (Other): All enrolled patients will have brain pulse monitoring
  Interventions: Device: Brain Pulse Oximeter

INTERVENTIONS:
Device: Brain Pulse Oximeter — Sensor is placed on the right and/or left forehead and maintained with an elasticized headband. The duration of monitoring will last for approximately 60 minutes per monitoring session to obtain sufficient data. Serial monitoring will occur on three consecutive days.

SUMMARY:
This is a study of adult patients with a severe and sudden brain injury who have a drain placed in their brain to measure pressure. The purpose of the study is to monitor the pressure in the brain using a monitor placed on the forehead, and compare this to a drain placed in the brain.

DETAILED DESCRIPTION:
The device is a non-invasive brain pulse oximeter. It uses red and near-infrared light and provides a signal which represents the change in blood volume associated with each heartbeat.

The brain signal allows a number of clinically important end-points to be determined, including brain blood flow, oxygen and pressure levels.

The T-Pot (US) Study will be undertaken in patients that require invasive brain monitoring.

The primary aim of the study is to assess the accuracy of the brain pulse oximeter compared with the traditional invasive intracranial pressure (ICP) monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult brain-injured patients who have undergone external ventricular drain insertion for cerebrospinal fluid drainage and invasive intracranial pressure monitoring as part of standard medical care
* 2. Adult brain-injured patients who have undergone external ventricular drain insertion for cerebrospinal fluid drainage and invasive intracranial pressure monitoring that have concomitant continuous electroencephalography (EEG) monitoring as part of standard medical care

Exclusion Criteria:

* 1. Inability to obtain the brain pulse oximeter signal from at least one brain hemisphere due to interface issue such as severe agitation, head dressing, severe skin or bone trauma, or skull removal preventing brain pulse detection for the initial monitoring session.

  a. Note: If unable to obtain brain pulse oximeter signal for subsequent monitoring sessions, the only the recordings that were obtained will be used for analysis
* 2. Hemodynamically unstable patients (defined as increasing vasopressors requirements)
* 3. Patients with unstable mechanical ventilation support defined as increasing fractional inspired oxygen (FiO2) requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Agreement of the brain oximeter levels compared with invasive ICP levels | Daily recordings for up to 30 days while the patient has an invasive ICP probe in situ
  Correlation of the optical signal waveforms with the invasive ICP waveforms and level

SECONDARY OUTCOMES:
Optical signal changes associated with periods of brain hypoxia and surrogate ICP waveform | Daily recordings for up to 30 days while the patient has an invasive ICP probe in situ
  Correlation of optical signal waveforms with clinical or other evidence of hypoxia
Optical signal changes associated with non-convulsive seizures via EEG monitoring (Alpha, Beta, Theta) | Daily recordings for up to 30 days while the patient has an invasive ICP probe in situ
  Correlation of optical signal waveforms with EEG monitoring (Alpha, Beta, Theta)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Hassett, DO, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Neurological Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No